CLINICAL TRIAL: NCT01959282
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Dose-response Study Evaluating the Efficacy and Safety of JNJ-54781532 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Safety and Effectiveness of JNJ-54781532 in Patients With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102640; 54781532UCO2001 (Other: Janssen Research & Development, LLC); 2013-000263-88 (EudraCT Number)
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, Ulcerative; JNJ-54781532; Moderate; Severe; Active
MeSH Terms: conditions — Colitis, Ulcerative; Lymphoma, Follicular; Motor Activity | interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (5):
- Placebo (Placebo Comparator): Participants will receive placebo once daily from Week 0 to Week 8. Participants in clinical response at Week 8 will continue to receive placebo through Week 32. Participants not in clinical response at Week 8 will receive treatment with 150 mg JNJ-54781532 orally once daily from Week 8 to Week 16. Participants who achieve a partial Mayo score response (ie, a change from baseline of ≥3 in the partial Mayo score) at Week 16 can continue receiving 150 mg JNJ-54781532 orally once daily through Week 32
  Interventions: Drug: Placebo; Drug: JNJ-54781532 150 mg once daily
- JNJ-54781532 25 mg once daily (Experimental): Participants will receive 25 mg of JNJ-54781532 once daily from Week 0 to Week 8. Participants in clinical response at Week 8 will continue to receive the same dosage through Week 32 and participants not in clinical response at Week 8 will continue to receive the same dosage through Week 16. At Week 16, participants who do not achieve a partial Mayo score response (ie, a change from baseline of ≥3 in the partial Mayo score) will be discontinued from study medication, and participants who achieve a partial Mayo score response at Week 16 can continue receiving JNJ 54781532 25 mg once daily through Week 32
  Interventions: Drug: JNJ-54781532 25 mg once daily
- JNJ-54781532 75 mg once daily (Experimental): Participants will receive 75 mg of JNJ-54781532 once daily from Week 0 to Week 8. Participants in clinical response at Week 8 will continue to receive the same dosage through Week 32 and participants not in clinical response at Week 8 will continue to receive the same dosage through Week 16. At Week 16, participants who do not achieve a partial Mayo score response (ie, a change from baseline of ≥3 in the partial Mayo score) will be discontinued from study medication, and participants who achieve a partial Mayo score response at Week 16 can continue receiving JNJ 54781532 75 mg once daily through Week 32
  Interventions: Drug: JNJ-54781532 75 mg once daily
- JNJ-54781532 150 mg once daily (Experimental): Participants will receive 150 mg of JNJ-54781532 once daily from Week 0 to Week 8. Participants in clinical response at Week 8 will continue to receive the same dosage through Week 32 and participants not in clinical response at Week 8 will continue to receive the same dosage through Week 16. At Week 16, participants who do not achieve a partial Mayo score response (ie, a change from baseline of ≥3 in the partial Mayo score) will be discontinued from study medication, and participants who achieve a partial Mayo score response at Week 16 can continue receiving JNJ 54781532 150 mg once daily through Week 32
  Interventions: Drug: JNJ-54781532 150 mg once daily
- JNJ-54781532 75 mg twice daily (Experimental): Participants will receive 75 mg of JNJ-54781532 twice daily from Week 0 to Week 8. Participants in clinical response at Week 8 will continue to receive the same dosage through Week 32 and participants not in clinical response at Week 8 will continue to receive the same dosage through Week 16. At Week 16, participants who do not achieve a partial Mayo score response (ie, a change from baseline of ≥3 in the partial Mayo score) will be discontinued from study medication, and participants who achieve a partial Mayo score response at Week 16 can continue receiving JNJ 54781532 75 mg twice daily through Week 32
  Interventions: Drug: JNJ-54781532 75 mg twice daily

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo once daily
  Arms: Placebo
Drug: JNJ-54781532 25 mg once daily — Participants will receive 25 mg of JNJ-54781532 once daily
  Other Names: ASP015K
  Arms: JNJ-54781532 25 mg once daily
Drug: JNJ-54781532 75 mg once daily — Participants will receive 75 mg of JNJ-54781532 once daily
  Other Names: ASP015K
  Arms: JNJ-54781532 75 mg once daily
Drug: JNJ-54781532 150 mg once daily — Participants will receive 150 mg of JNJ-54781532 once daily
  Other Names: ASP015K
  Arms: JNJ-54781532 150 mg once daily; Placebo
Drug: JNJ-54781532 75 mg twice daily — Participants will receive 75 mg of JNJ-54781532 twice daily
  Other Names: ASP015K
  Arms: JNJ-54781532 75 mg twice daily

SUMMARY:
The purpose of the study is to evaluate dose response of JNJ-54781532 in participants with moderately to severely active ulcerative colitis (UC).

DETAILED DESCRIPTION:
This is a Phase 2b, multicenter, randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study), parallel-group (each group of participants will be treated at the same time), dose-response study (a study to evaluate response to different dosages of study medication) of oral tablets of JNJ-54781532 in adult participants with moderately to severely active UC. Approximately 220 participants will be randomized in a 1:1:1:1:1 ratio to 1 of 5 treatment groups at Week 0 (placebo; JNJ-54781532 25 mg once daily; JNJ-54781532 75 mg once daily; JNJ-54781532 150 mg once daily; and JNJ-54781532 75 mg twice daily) to receive their randomized dosage of study medication through Week 8 and will be assessed for clinical response at Week 8. Participants who achieve clinical response at Week 8 will continue to receive their original randomized dosage of study medication through Week 32. Participants who do not achieve clinical response at Week 8 will be treated as follows: participants originally randomized to placebo will receive JNJ-54781532 150 mg once daily through Week 16; participants originally randomized to JNJ-54781532 will continue to receive their original randomized dosage of JNJ-54781532 through Week 16. Participants who were not in clinical response at Week 8 and do not achieve a partial Mayo score response (a decrease from baseline in the partial Mayo score by ≥3 points) at Week 16 will be discontinued from study medication; and those who achieve a partial Mayo score response at Week 16 can continue receiving JNJ 54781532 through Week 32. Participants will be evaluated for safety (adverse events) up to Week 36 (ie, 4 weeks after the last dose of study medication). The maximum study duration for each participant will be approximately 44 weeks (including maximum screening period).

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of ulcerative colitis (UC) at least 3 months prior to screening
* Have moderately to severely active UC, defined as a baseline (Week 0) Mayo score of 6 to 12; including an endoscopy sub score greater than or equal to 2 as determined by a central read of the video endoscopy
* Current treatment with oral corticosteroids or have a history of failure to respond to, or tolerate, at least 1 of the following therapies oral corticosteroids (including budesonide), 6-mercaptopurine (6-MP), azathioprine (AZA), or anti- tumor necrosis factor therapy or be corticosteroid dependent (ie, an inability to successfully taper corticosteroids without a return of the symptoms of UC)
* Must discontinue 6-MP/AZA for at least 1 week before the first dose of study medication

Exclusion Criteria:

* At imminent risk for colectomy
* Have ulcerative colitis limited to the rectum only or to less than 20 centimeter of the colon
* Presence of a stoma
* Presence or history of a fistula
* History or current diagnosis of active or latent tuberculosis; human immunodeficiency virus; hepatitis C virus or hepatitis B virus infection; have had more than 1 herpes zoster infection or have had any diagnosis of disseminated herpes zoster
* Previous treatment with a janus kinase inhibitor (eg, tofacitinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2015-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Mayo score at Week 8 | Week 8
  The Mayo score is the primary tool for assessing ulcerative colitis activity. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, findings of endoscopy, and physician's global assessment) which range from 0 to 3. The Mayo score is calculated as the sum of these 4 subscores and can range between 0 and 12. A score of 3 to 5 points indicates mildly active disease; a score of 6 to 10 indicates moderately active disease; and a score of 11 to 12 indicates severe disease.

SECONDARY OUTCOMES:
Number of participants with clinical response at Week 8 | Week 8
  Clinical response is defined as a decrease from baseline in the Mayo score by ≥30% and ≥3 points, with either a decrease from baseline in the rectal bleeding subscore of ≥1 or a rectal bleeding subscore of 0 or 1.
Number of participants with clinical remission at Week 8 | Week 8
  Clinical remission is defined as a Mayo score ≤2 points, with no individual subscore >1.
Number of participants with mucosal healing at Week 8 | Week 8
  Mucosal healing is an improvement in the endoscopic appearance of the mucosa. An endoscopy subscore of the Mayo score of 0 or 1.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (97):
- United States (15):
  - La Jolla, California
  - Thornton, Colorado
  - Ann Arbor, Michigan
  - Tupelo, Mississippi
  - Egg Harbor, New Jersey
  - Salisbury, North Carolina
  - Cleveland, Ohio
  - Lima, Ohio
  - Norman, Oklahoma
  - Germantown, Tennessee
  - Nashville, Tennessee
  - San Antonio, Texas
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Seattle, Washington
- Australia (8):
  - Bankstown
  - Bedford
  - Concord
  - Herston
  - Launceston
  - Melbourne
  - Penrith
  - South Brisbane
- Belgium (4):
  - Brussels
  - Ghent
  - Kortrijk
  - Leuven
- Bulgaria (3):
  - Pleven
  - Sofia
  - Varna
- Canada (8):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Greater Sudbury, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (3):
  - Lille
  - Paris
  - Pessac
- Germany (12):
  - Berlin
  - Essen
  - Frankfurt A. M.
  - Hanover
  - Heidelberg
  - Herne
  - Jena
  - Kiel
  - Magdeburg
  - Münster
  - Neustadt
  - Stade
- Hungary (4):
  - Békéscsaba
  - Budapest
  - Mosonmagyaróvár
  - Szekszárd
- Israel (6):
  - Hadera
  - Haifa
  - Jerusalem
  - Nazareth
  - Ramat Gan
  - Rehovot
- Netherlands (4):
  - Amsterdam
  - Amsterdam-Zuidoost
  - Maastricht
  - Rotterdam
- Poland (4):
  - Elblag
  - Lodz
  - Sopot
  - Warsaw
- Romania (4):
  - Bucharest
  - Constanța
  - Iași
  - Timișoara
- Russia (10):
  - Kazan’
  - Nizny Novgorod
  - Novosibirsk
  - Omsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Stavropol
  - Ufa
  - Yaroslavl
- Ukraine (12):
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Odesa
  - Ternopil
  - Uzhhorod
  - Vinnitsa
  - Zaporizhzhia
  - Zhaporozhia 69104

REFERENCES:
- [Derived] Li K, Strauss R, Marano C, Greenbaum LE, Friedman JR, Peyrin-Biroulet L, Brodmerkel C, De Hertogh G. A Simplified Definition of Histologic Improvement in Ulcerative Colitis and its Association With Disease Outcomes up to 30 Weeks from Initiation of Therapy: Post Hoc Analysis of Three Clinical Trials. J Crohns Colitis. 2019 Aug 14;13(8):1025-1035. doi: 10.1093/ecco-jcc/jjz022. PMID 30721964
- [Derived] Sands BE, Sandborn WJ, Feagan BG, Lichtenstein GR, Zhang H, Strauss R, Szapary P, Johanns J, Panes J, Vermeire S, O'Brien CD, Yang Z, Bertelsen K, Marano C; Peficitinib-UC Study Group. Peficitinib, an Oral Janus Kinase Inhibitor, in Moderate-to-severe Ulcerative Colitis: Results From a Randomised, Phase 2 Study. J Crohns Colitis. 2018 Nov 9;12(10):1158-1169. doi: 10.1093/ecco-jcc/jjy085. PMID 29917064
- See also: Related Info — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-000263-88/results